CLINICAL TRIAL: NCT02704988
Title: Clinical Trial Comparing Carnoy's and GEWF Solutions for Lymph Node Clearing Technique in Colorectal Cancer
Brief Title: Clinical Trial Comparing Carnoy's and GEWF Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HMV-CRC1
Record Dates: First submitted 2016-02-22; First posted 2016-03-10 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Lymph Node Metastasis; Colorectal Cancer
MeSH Terms: conditions — Lymphatic Metastasis; Colorectal Neoplasms | interventions — gewf solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Colon Cancer - Carnoy (Active Comparator): (1) just after the surgical resection each specimen is fixed by formaldehyde; (2) lymph node harvesting is performed by a manual technique of vision and palpation; (3) lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy; (4) the surgical specimen is submitted to re-fixation with Carnoy solution and another lymph node harvesting by manual technique of vision and palpation; (5) additional lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy.
  Interventions: Procedure: Carnoy Solution
- Colon Cancer - GEWF (Active Comparator): (1) just after the surgical resection each specimen is fixed by formaldehyde; (2) lymph node harvesting is performed by a manual technique of vision and palpation; (3) lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy; (4) the surgical specimen is submitted to re-fixation with GEWF solution and another lymph node harvesting by manual technique of vision and palpation; (5) additional lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy.
  Interventions: Procedure: GEWF Solution
- Rectal Cancer - Carnoy (Active Comparator): (1) just after the surgical resection each specimen is fixed by formaldehyde; (2) lymph node harvesting is performed by a manual technique of vision and palpation; (3) lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy; (4) the surgical specimen is submitted to re-fixation with Carnoy solution and another lymph node harvesting by manual technique of vision and palpation; (5) additional lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy.
  Interventions: Procedure: Carnoy Solution
- Rectal Cancer - GEWF (Active Comparator): (1) just after the surgical resection each specimen is fixed by formaldehyde; (2) lymph node harvesting is performed by a manual technique of vision and palpation; (3) lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy; (4) the surgical specimen is submitted to re-fixation with GEWF solution and another lymph node harvesting by manual technique of vision and palpation; (5) additional lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy.
  Interventions: Procedure: GEWF Solution

INTERVENTIONS:
Procedure: Carnoy Solution — The subjects in this group will undergo intervention by having surgery (colorectal cancer resection) and lymph node clearing technique with Carnoy solution
  Arms: Colon Cancer - Carnoy; Rectal Cancer - Carnoy
Procedure: GEWF Solution — The subjects in this group will undergo intervention by having surgery (colorectal cancer resection) and lymph node clearing technique with GEWF solution
  Arms: Colon Cancer - GEWF; Rectal Cancer - GEWF

SUMMARY:
Regional lymph node metastasis is a major determinant of local recurrence and overall survival rates in patients with colorectal cancer. Because of the poor prognosis associated with the presence of lymph node metastasis, stage III colorectal cancer patients should receive adjuvant treatment with chemo and / or radiation therapy according to the site of tumor. Several authors have investigated the use of revealing solutions for lymph node clearance in colorectal cancer. Most studies comparing conventional histopathological specimen examination to any lymph node clearing technique showed that the use of revealing solutions increases the mean number of lymph nodes harvested, usually in a statistically significant manner. It is still controversial the impact of the use of revealing solutions for upstaging of lymph node status and consequently for the indication for adjuvant therapy. Therefore will be conducted a randomized clinical trial to compares the performance of GEWF and Carnoy solutions for the histopathological examination of patients with colorectal cancer. The aim of this study is to determine the lymph node revealing solution with the best performance (increase in the mean number of lymph node harvested and lymph node upstaging) in patients with colorectal cancer.

DETAILED DESCRIPTION:
Colorectal adenocarcinoma patients, consecutively submitted to surgical treatment performed by colorectal surgeons with more than 10 years of professional experience at Hospital Moinhos de Vento (Porto Alegre, Brazil), will have their surgical specimens subjected to conventional anatomopathological examination for the analysis of the lymph nodes (visual and palpation) performed by a highly qualified pathology technician in lymph node clearing technique. The lymph nodes identified in this preliminary examination will be counted and submitted to pathologic examination with hematoxylin and eosin staining for lymph node metastasis by a pathologist with over 10 years of experience. Upon completing this procedure with the patients with colon cancer, those with rectal cancer will be randomized and have their surgical specimens submitted to the lymph node clearing technique with Carnoy's or GEWF solutions, according to the groups below.

1. Colon Cancer Group - Carnoy Procedure: The surgical resection specimen will be embedded in a plastic container with 1000 ml of Carnoy solution for 24 to 48 hours. Carnoy's solution is a fixative composed of 60% ethanol, 30% chloroform and 10% glacial acetic acid. Following, a technician in pathological macroscopy with 10 years of experience will perform a visual and manual assessment of additional lymph nodes for 60 minutes. Each additional lymph node identified will be entirely or partially embedded, depending on the size, in paraffin and subsequently stained with hematoxylin-eosin.The microscopic examination of the slides obtained from the anatomopathological examination with Carnoy's solution will be performed by two pathologists with seven and 25 years of experience, respectively, both with wide experience in lymph node clearing technique.
2. Colon Cancer Group - GEWF Procedure: The surgical resection specimen will be embedded in a plastic container with 1000 ml of GEWF solution for 24 to 48 hours. GEWF solution is a fixative composed of 62.5% ethanol, 21.25% distilled water, 10% formaldehyde and 6.25% glacial acetic acid. Following, a technician in pathological macroscopy with 10 years of experience will perform a visual and manual assessment of additional lymph nodes for 60 minutes. Each additional lymph node identified will be entirely or partially embedded, depending on the size, in paraffin and subsequently stained with hematoxylin-eosin.

   The microscopic examination of the slides obtained from the anatomopathological examination with Carnoy's solution will be performed by two pathologists with seven and 25 years of experience, respectively, both with wide experience in lymph node clearing technique.
3. Rectal Cancer Group - Carnoy Procedure: The surgical resection specimen will be embedded in a plastic container with 1000 ml of Carnoy solution for 24 to 48 hours. Carnoy's solution is a fixative composed of 60% ethanol, 30% chloroform and 10% glacial acetic acid. Following, a technician in pathological macroscopy with 10 years of experience will perform a visual and manual assessment of additional lymph nodes for 60 minutes. Each additional lymph node identified will be entirely or partially embedded, depending on the size, in paraffin and subsequently stained with hematoxylin-eosin.The microscopic examination of the slides obtained from the anatomopathological examination with Carnoy's solution will be performed by two pathologists with seven and 25 years of experience, respectively, both with wide experience in lymph node clearing technique.
4. Rectal Cancer Group - GEWF Procedure: The surgical resection specimen will be embedded in a plastic container with 1000 ml of GEWF solution for 24 to 48 hours. GEWF solution is a fixative composed of 62.5% ethanol, 21.25% distilled water, 10% formaldehyde and 6.25% glacial acetic acid. Following, a technician in pathological macroscopy with 10 years of experience will perform a visual and manual assessment of additional lymph nodes for 60 minutes. Each additional lymph node identified will be entirely or partially embedded, depending on the size, in paraffin and subsequently stained with hematoxylin-eosin. The microscopic examination of the slides obtained from the anatomopathological examination with Carnoy's solution will be performed by two pathologists with seven and 25 years of experience, respectively, both with wide experience in lymph node clearing technique.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma
* Voluntary agreement of the patient to participate in research
* Voluntary agreement of the surgeon to participate in research

Exclusion Criteria:

* Absence of accurate histopathological data
* Unplanned extended resection
* Synchronous colorectal cancer
* Inflammatory bowel disease
* Extended lymphadenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2015-03; Primary Completion 2018-06 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Increased lymph node sample | 1 week
  Additional number (unit measure) of lymph nodes identified by the lymph node clearing technique (visual and manual examination with Carnoy's or GEWF solutions) compared to the initial number (unit measure) of lymph nodes identified by the conventional technique (visual and manual examination with formaldehyde).

SECONDARY OUTCOMES:
Additional lymph node metastases | 1 week
  Presence of metastases in the additional lymph nodes harvested
Change of lymph node staging | 1 week
  Increase of lymph node staging status (migration from N classification to higher staging), according to the 7th edition of the American Joint Committee on Cancer, with the lymph node clearing technique (visual and manual examination with Carnoy's or GEWF solutions) compared to the initial lymph node staging by the conventional technique (visual and manual examination with formaldehyde).
Indication for adjuvant treatment | 1 month
  Patient (unit measure) who had indication for adjuvant treatment (chemotherapy, radiotherapy or combined chemoradiotharepy) to treat colorectal cancer due to the outcome changes of the lymph node staging after using the lymph node clearing technique (visual and manual examination with Carnoy's or GEWF solutions).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio N Kalil, MD, PhD, Study Chair — Federal University of Health Science of Porto Alegre
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No